CLINICAL TRIAL: NCT00958282
Title: Lisdexamfetamine Treatment for Cocaine Dependence
Brief Title: Treatment of Cocaine Dependence With Lisdexamfetamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0812M54801; DA023548 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-08

CONDITIONS: Cocaine Dependence
Keywords: cocaine; treatment; lisdexamfetamine; dependence; addiction; crack
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Lisdexamfetamine Dimesylate; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lisdexamfetamine/Behavior Therapy (Active Comparator): lisdexamfetamine 70mg/day plus Behavior Therapy
  Interventions: Drug: lisdexamfetamine/Behavior Therapy
- placebo (Placebo Comparator): Placebo Comparator once per day
  Interventions: Other: placebo

INTERVENTIONS:
Drug: lisdexamfetamine/Behavior Therapy
  Arms: lisdexamfetamine/Behavior Therapy
Other: placebo
  Arms: placebo

SUMMARY:
This protocol is a 2-group double-blind placebo-controlled outpatient study investigating lisdexamfetamine for treatment of cocaine dependence. The investigators plan to enroll 100 subjects in a 14-week trial. The primary objectives will determine changes in cocaine use and secondary objectives will be cocaine craving and impulsivity.

DETAILED DESCRIPTION:
This 2-group, double-blind, placebo-controlled, 14-week study (N=100) will investigate the efficacy of cognitive behavioral therapy plus lisdexamfetamine vs. placebo to treat cocaine dependence. We hypothesize that lisdexamfetamine will reduce cocaine use (primary outcome), as well as cocaine craving and impulsivity (secondary outcomes) vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must:

  1. Be treatment-seeking males or females between 18 and 65 years-of-age;
  2. Understand the study procedures and provide written informed consent;
  3. Be judged by the examining physician to be in generally good health with the exception of health problems related to acute drug use;
  4. Meet DSM-IV criteria for cocaine-dependence.

Exclusion Criteria:

* Exclusion criteria include:

  1. DSM-IV diagnoses for current psychotic disorders, mood disorders (except substance-induced depression), anxiety disorders, ADHD, and other current substance dependence (except marijuana and nicotine dependence); subjects may not have physiological dependence upon alcohol requiring medical detoxification;
  2. Current use of any prescription medications;
  3. Females currently pregnant or nursing;
  4. Current elevation of liver enzyme levels above twice normal limits;
  5. Existing cardiovascular disease as determined by physician, EKG evaluation;
  6. History of significant acute or chronic physical illness precluding participation;
  7. History of hyperthyroidism, glaucoma, or seizures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Mooney, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Ambulatory Research Center/Fairview University Psychiatry Dept, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisdexamfetamine: lisdexamfetamine 70mg/day
  lisdexamfetamine
  cognitive behavioral therapy
- Placebo: Placebo Comparator once per day
  placebo
  cognitive behavioral therapy
Period: Overall Study
Arm/Group | Lisdexamfetamine | Placebo
Started | 22 | 21
Completed | 12 | 15
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (5.9) | 46.4 (10) | 46.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 18 | 17 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 14 | 12 | 26
  White | 8 | 4 | 12
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Cocaine-positive Urine Results
Description: At each visit, subjects provided urine samples, which were analyzed for benzoylecgonine (BE; a cocaine metabolite). BE was assessed semi-quantitatively using the PROFILE® -V MEDTOXScan® Drugs of Abuse Test System, with cocaine positive tests equaling or exceeding 150 ng/mL.
Time Frame: 14 Weeks
Measure: Mean (Standard Deviation); unit: percentage of BE urine tests
Arm/Group | Lisdexamfetamine | Placebo
Number analyzed (Participants) | 22 | 21
percentage of BE urine tests | 86.5 (.5) | 92.4 (.5)

2. Secondary Outcome: Drug Craving
Description: On a weekly basis, patients completed measures of cocaine craving using the Minnesota Cocaine Craving Scale.
  The Minnesota Cocaine Craving Scale is a self report questionnaire and ranges from 0 to 100, 0 being "very little" to 100 being "very much".
Time Frame: 14 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lisdexamfetamine | Placebo
Number analyzed (Participants) | 22 | 21
units on a scale | 17.5 (3.30) | 28.7 (3.21)

ADVERSE EVENTS:
Groups:
- Lisdexamfetamine/Behavior Therapy: lisdexamfetamine 70mg/day plus Behavior Therapy
  lisdexamfetamine/Behavior Therapy
- Placebo: Placebo Comparator once per day
  placebo
Arm/Group | Lisdexamfetamine/Behavior Therapy | Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine/Behavior Therapy (N=22) | Placebo (N=21)
Angina (Cardiac disorders) | 1 (1) | 0 (0) — A patient was hospitalized for chest pain and diagnosed with angina that was possibly related to the study drug. He did not continue in the study. He was assigned to the LDX condition.
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) — A subject was hospitalized with psychosis (assigned to the placebo condition). She had apparently binged on cocaine prior to her psychotic episode. In addition she failed to reveal to study staff that she was diagnosed with schizoaffective disorder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes